CLINICAL TRIAL: NCT06307327
Title: A Comparative Study on the Evaluation Consistency Between the New Type and the Traditional Grade of Radioactive Oropharyngeal Mucositis and the Exploration of Blood Markers
Brief Title: Comparative Study of New Classification and Traditional Classification of Radioactive Oropharyngeal Mucositis
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-098
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Radiation-Induced Mucositis
Keywords: Radiation oropharyngeal mucositis; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiation oropharyngeal mucositis is one of the most painful side effects of radiotherapy in patients with head and neck tumors. However, the traditional radioactive oropharyngeal mucositis grading system has the problem of poor evaluation consistency. To solve this problem, we innovatively classify radiation oropharyngeal mucositis into four types according to the four-stage histopathological changes of acute radiation injury: (1) congestive; (2) Scattered erosion type; (3) Fusion erosion type; (4) Ulcer type. We intend to conduct a multicenter observational cohort study to compare the consistency of different physicians in the assessment of radiation oropharyngeal mucositis with new and traditional classifications, and to explore changes in blood markers of different types of oropharyngeal mucositis using clinical residual blood samples.

DETAILED DESCRIPTION:
Since this is an observational study, no additional visits, laboratory analyses, or evaluations beyond the routine clinical practice requirements are necessary. Patients must sign the latest informed consent form (ICF) approved by the ethics committee before data collection is carried out. After obtaining the patient's consent, clinical routine diagnosis and treatment information will be collected.

The study is divided into three parts. The first part compares the consistency of results among different methods used to assess mucositis. The research process involves having different doctors assess the same patient at the same stage using a specific grading method three times, and taking the results of more than two of these assessments as the internal unified results of that grading method (each patient can be assessed and data recorded every 1-2 weeks during radiotherapy). After obtaining the internal unified results of the three mucositis grading methods, the consistency of results among different methods used for assessment is compared.

The second part first determines the internal consistency of doctor evaluations for four methods (the traditional three mucositis grading methods and the new classification method), and then uses the consistency results of each method to compare the stability of the assessments. The research process involves having different doctors assess the same patient at the same stage using a specific method three times. Each patient can be assessed and data recorded every 1-2 weeks during radiotherapy. The consistency of evaluations among different doctors for this method is obtained. Finally, this consistency is used to compare the stability of the assessments between different methods.

The third part compares the consistency of results between the assessment using the new mucositis classification method and the patient's self-assessment. The research process involves having different doctors assess the same patient at the same stage using the new classification method three times, and taking the results of more than two of these assessments as the internal unified result of the new classification method (each patient can be assessed and data recorded every 1-2 weeks during radiotherapy). After obtaining the internal unified results of the new classification method and the patient's self-assessment results, the consistency of results between using the new classification method and the patient's self-assessment is compared.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign informed consent;
* Age 18 or older on the date of signing the informed consent;
* Histologically confirmed head and neck tumor, radiotherapy or chemoradiotherapy.

Exclusion Criteria:

* They also have other uncontrolled serious medical conditions, such as unstable heart disease requiring treatment, poorly controlled diabetes (fasting blood glucose > 1.5× the upper limit of normal), mental illness, and a history of severe allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects in this study were head and neck tumor patients receiving radiotherapy
Sampling Method: Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Inter-rater consistency among doctors | Through study completion, up to 3 years
  Different physician assessments of agreement (percentage) were directly compared between the new and traditional classifications. Consistency refers to the proportion of assessments made by two doctors that are the same.

SECONDARY OUTCOMES:
Consistency in assessment between doctors and patients | Through study completion, up to 3 years
  In the new classification, the consistency (percentage) of assessment between doctors and patients was compared. Consistency refers to the proportion of times where the assessments made by the two doctors were the same.
The assessment period | Through study completion, up to 3 years
  The assessment times used respectively for different assessment methods
the satisfaction of patients | Through study completion, up to 3 years
  the satisfaction of patients
the satisfaction of doctors | Through study completion, up to 3 years
  the satisfaction of doctors

OTHER OUTCOMES:
Exploration of blood biomarkers related to the classification of radioactive oropharyngeal mucositis | Through study completion, up to 3 years
  Exploration of blood biomarkers related to the classification of radioactive oropharyngeal mucositis

CONTACTS AND LOCATIONS:
Overall Officials: Jian Guan, M.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (4):
- China (4):
  - Southern medical university, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Jieyang people's hospital, Jieyang, Guangdong
  - Meizhou People's Hospital, Meizhou Academy of Medical Sciences Meizhou, Meizhou, Guangdong

IPD SHARING:
Plan to Share IPD: No